CLINICAL TRIAL: NCT00128102
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial of Oral Suberoylanilide Hydroxamic Acid (Vorinostat, MK-0683) in Patients With Advanced Malignant Pleural Mesothelioma Previously Treated With Systemic Chemotherapy
Brief Title: Suberoylanilide Hydroxamic Acid (Vorinostat, MK-0683) Versus Placebo in Advanced Malignant Pleural Mesothelioma (MK-0683-014)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0683-014; 2005_010 (Other: Merck registration number); CTRI/2009/091/000146 (Registry Identifier: CTRI); MK-0683-014 (Other: Merck); NCT00265577 (obsolete NCT alias); NCT00290784 (obsolete NCT alias)
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Mesothelioma; Lung Cancer
Keywords: Advanced malignant pleural mesothelioma
MeSH Terms: conditions — Mesothelioma; Lung Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vorinostat (Experimental): Vorinostat three 100 mg capsules twice daily for 3 consecutive days of treatment followed by 4 days of rest repeated weekly, in 21-day cycles. Treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Vorinostat
- Placebo (Placebo Comparator): Placebo capsules twice daily for 3 consecutive days of treatment followed by 4 days of rest repeated weekly, in 21-day cycles. Treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vorinostat — Vorinostat 100 mg oral capsules
  Other Names: MK-0683; Zolinza
  Arms: Vorinostat
Drug: Placebo — Vorinostat-matching placebo oral capsules
  Arms: Placebo

SUMMARY:
The goal of this study is to assess the efficacy and safety of an oral investigational drug suberoylanilide hydroxamic acid (vorinostat, MK-0683) compared to placebo, in the treatment of participants with advanced malignant pleural mesothelioma who have failed at least one prior chemotherapy regimen. The primary hypotheses are the following: (1) vorinostat improves overall survival (OS) compared to placebo (2) vorinostat is generally safe and well tolerated.

DETAILED DESCRIPTION:
Treatment Extension Phase: Participants in this study will be eligible to enroll in an open-label treatment extension phase if they: a) were originally randomized to the vorinostat arm and have not experienced disease progression; b) were randomized to the placebo arm and meet the "Extension Phase Inclusion Criteria for Participants in the Placebo Arm" below; or c) were originally randomized to the vorinostat arm and discontinued study therapy for reasons other than progression and the investigator believes that it is in the participant's best interest to resume vorinostat treatment.

As specified by the protocol, based on planned extension phase inclusion criteria and pre-specified primary outcome analyses requirements, the extension phase of this study was not conducted.

ELIGIBILITY:
Inclusion Criteria :

* 18 years or older with confirmed diagnosis of malignant pleural mesothelioma
* In countries where pemetrexed is an approved mesothelioma treatment, the participant's disease has progressed or relapsed following treatment with at least one prior chemotherapy regimen with pemetrexed and either cisplatin or carboplatin OR in countries where pemetrexed is not approved for mesothelioma, the participant's disease has progressed or relapsed following treatment with at least one prior chemotherapy regimen OR pemetrexed is not the preferred therapy for the participant and the participant's disease has progressed or relapsed following treatment with at least one prior chemotherapy regimen
* Received no more than 2 prior systemic therapy regimens
* Karnofsky performance scale status of ≥70
* Has adequate bone marrow, liver, and kidney function and adequate coagulation (per prespecified laboratory values)

Extension Phase Inclusion Criteria:

* Participants who are receiving treatment with vorinostat and have not experienced progression of mesothelioma
* Randomized to the placebo arm and: 1) have a Karnofsky performance scale status of ≥70; and 2) have adequate bone marrow, liver, and kidney function and adequate coagulation (per prespecified laboratory values)
* Randomized to vorinostat and have discontinued study therapy for reasons other than progression of mesothelioma, if the investigator is of the opinion that the potential benefit outweighs potential risks associated with using vorinostat

Exclusion Criteria:

* Has an active infection for which they received treatment with intravenous antibiotic, antiviral, or antifungal medications within 2 weeks of the start of study drug.
* Has a "currently active" second malignancy; a malignancy is not considered "currently active" if participants have completed therapy for the second malignancy and are disease free from prior malignancies for >5 years
* Has uncontrolled brain metastases
* Has a known human immunodeficiency virus (HIV) infection or HIV-related malignancy
* Is pregnant or breast feeding
* Has a history of gastrointestinal surgery or other procedures that might interfere with the absorption or swallowing of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2005-06-30 (Actual); Primary Completion 2011-07-15 (Actual); Study Completion 2011-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Krug LM, Kindler HL, Calvert H, Manegold C, Tsao AS, Fennell D, Ohman R, Plummer R, Eberhardt WE, Fukuoka K, Gaafar RM, Lafitte JJ, Hillerdal G, Chu Q, Buikhuisen WA, Lubiniecki GM, Sun X, Smith M, Baas P. Vorinostat in patients with advanced malignant pleural mesothelioma who have progressed on previous chemotherapy (VANTAGE-014): a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Oncol. 2015 Apr;16(4):447-56. doi: 10.1016/S1470-2045(15)70056-2. Epub 2015 Mar 20. PMID 25800891

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat: Vorinostat three 100 mg capsules twice daily for 3 consecutive days of treatment followed by 4 days of rest repeated weekly, in 21-day cycles. Treatment continued until disease progression or unacceptable toxicity.
- Placebo: Placebo capsules twice daily for 3 consecutive days of treatment followed by 4 days of rest repeated weekly, in 21-day cycles. Treatment continued until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Vorinostat | Placebo
Started | 329 | 332
Treated | 329 | 329
Completed | 1 | 0
Not Completed | 328 | 332
Not completed — Site Discontinued | 3 | 6
Not completed — Other | 0 | 1
Not completed — Progressive Disease | 255 | 285
Not completed — Adverse Event | 34 | 11
Not completed — Death | 12 | 13
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 19 | 11
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat | Placebo | Total
Number analyzed (Participants) | 329 | 332 | 661
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (9.5) | 64.4 (9.3) | 64.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 62 | 108
  Male | 283 | 270 | 553

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of final analysis were censored at the date of the last follow up. The final analysis for OS was planned and performed at the time of the protocol pre-specified final statistical analysis with a data cut-off of 15-July-2011. OS analysis is reported here for all randomized participants.
Time Frame: Up to ~72 months (through pre-specified final statistical analysis cut-off date of 15-July-2011)
Population: All participants randomized to a study arm.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 329 | 332
Weeks | 30.7 [26.71 to 36.14] | 27.1 [23.14 to 31.86]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p = 0.858, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.83 to 1.17]

2. Primary Outcome: Number of Participants Who Experienced Adverse Events (AEs) Characterized as Grade 3 or Grade 4 According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with the use of the Sponsor's product whether or not considered related to the use of the product. Any worsening of a pre-existing condition which is temporally associated with the use of the Sponsor's product is also an AE. Reporting of AEs per NCI CTCAE is based on 5 grades of severity; Grade 1 (mild; no treatment needed), Grade 2 (moderate; minimal treatment needed), Grade 3 (severe, not life threatening; hospitalization needed), Grade 4 (life threatening; urgent treatment needed) and Grade 5 (death).The final analysis for Grade 3 or 4 AEs was planned and performed at the time of the protocol pre-specified final statistical analysis with a data cut-off of 15-July-2011. Per protocol number of participants who experienced Grade 3/4 AEs per NCI CTCAE is reported here for all randomized participants who received ≥1 dose of study treatment.
Time Frame: Up to ~72 months (through pre-specified final statistical analysis cut-off date of 15-July-2011)
Population: All participants randomized to a study arm who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 329 | 329
Participants | 165 | 146

3. Primary Outcome: Number of Participants Who Experienced an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with the use of the Sponsor's product whether or not considered related to the use of the product. Any worsening of a pre-existing condition which is temporally associated with the use of the Sponsor's product is also an AE. The final analysis for participants who experienced an AE was planned and performed at the time of the protocol pre-specified final statistical analysis with a data cut-off of 15-July-2011. Per protocol number of participants who experienced an AE is reported here for all randomized participants who received ≥1 dose of study treatment.
Time Frame: Up to ~72 months (through pre-specified final statistical analysis cut-off date of 15-July-2011)
Population: All participants randomized to a study arm who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 329 | 329
Participants | 327 | 311

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with the use of the Sponsor's product whether or not considered related to the use of the product. Any worsening of a pre-existing condition which is temporally associated with the use of the Sponsor's product is also an AE. The final analysis for participants who discontinued study treatment due to an AE was planned and performed at the time of the protocol pre-specified final statistical analysis with a data cut-off of 15-July-2011. Per protocol number of participants who discontinued study treatment due to an AE is reported here for all randomized participants who received ≥1 dose of study treatment. As specified by the protocol, participants who discontinued study treatment due to an AE remained on study until investigator notification to discontinue.
Time Frame: Up to ~72 months (through pre-specified final statistical analysis cut-off date of 15-July-2011)
Population: All participants randomized to a study arm who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 329 | 329
Participants | 60 | 49

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per meso-modified-Response Evaluation Criteria in Solid Tumors (Meso-modified RECIST) based on independent radiology review or death due to any cause, whichever occurred first. Meso-modified RECIST was created and validated for disease measurement in pleural mesothelioma. Per meso-modified RECIST, PD was defined as ≥20% increase in the total tumor measurement over the nadir measurement or the appearance of ≥1 new lesions. The final analysis for PFS per Meso-modified RECIST by independent radiology review was planned and performed at the time of the protocol pre-specified final statistical analysis with a data cut-off of 15-July-2011. PFS analysis per Meso-modified RECIST by independent radiology review is reported here for all randomized participants.
Time Frame: Up to ~72 months (through pre-specified final statistical analysis cut-off date of 15-July-2011)
Population: All participants randomized to a study arm.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 329 | 332
Weeks | 6.3 [6.1 to 7.1] | 6.1 [6.0 to 6.1]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p < 0.001, Likelihood Based Score Test; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.63 to 0.88]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis population who had a complete response (CR: disappearance of all target lesions with no evidence of tumor elsewhere) or a partial response (PR: ≥30% reduction in the total tumor measurement) per Meso-modified RECIST based on independent radiology review. Meso-modified RECIST was created and validated for disease measurement in pleural mesothelioma. The final analysis for ORR per Meso-modified RECIST by independent radiology review was planned and performed at the time of the protocol pre-specified final statistical analysis with a data cut-off of 15-July-2011. Per protocol percentage of participants who had a CR or a PR per Meso-modified RECIST by independent radiology review is reported here as the ORR for all randomized participants who had valid baseline data for ORR analysis available.
Time Frame: Up to ~72 months (through pre-specified final statistical analysis cut-off date of 15-July-2011)
Population: All participants randomized to a study arm who had valid baseline data for ORR analysis available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 318 | 323
Percentage of Participants | 0.63 [0.08 to 2.25] | 0.31 [0.01 to 1.71]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p = 0.621, Fisher Exact; Difference in Percentage = 0.3, 95% CI 2-sided [-1.18 to 1.97]

7. Secondary Outcome: Percent Change From Baseline in Lung Cancer Symptom Scale, Modified for Mesothelioma (LCSS-Meso) Dyspnea Score at Week 12
Description: LCSS-Meso provides participant-reported outcome measures of symptom burden and quality of life. LCSS-Meso includes the disease-related item dyspnea or shortness of breath. The LCSS-Meso item dyspnea is measured on a visual analog scale (VAS) using 100 mm and assigned an individual score based on symptom intensity. Dyspnea VAS score ranges from 0 mm (lowest; no dyspnea) to 100 mm (highest; worst dyspnea). Higher scores indicate dyspnea worsening. Baseline measurement was taken before treatment initiation. Per protocol percent change in the LCSS-Meso dyspnea score from baseline to Week 12 post treatment initiation (percent change calculated: [Week 12 - Baseline]/Baseline*100)] is reported here for all randomized participants who had a valid baseline and ≥1 post-baseline value for the LCSS-Meso dyspnea score available.
Time Frame: Baseline, Week 12
Population: All participants randomized to a study arm who had a valid baseline and ≥1 post-baseline value for the LCSS-Meso dyspnea score available.
Measure: Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 299 | 299
Percent Change | 141.8 [72.9 to 210.8] | 174.7 [40.4 to 308.9]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p = 0.259, Longitudinal Model; Difference in Percent Change = -52.4, 95% CI 2-sided [-143.5 to 38.6]

8. Secondary Outcome: Percentage of Participants With ≥50% Change Together With a >10 mm Change From Baseline in the LCSS-Meso Dyspnea Score at Week 12
Description: LCSS-Meso provides participant-reported outcome measures of symptom burden and quality of life. LCSS-Meso includes the disease-related item dyspnea or shortness of breath. The LCSS-Meso item dyspnea is measured on a visual analog scale (VAS) using 100 mm and assigned an individual score based on symptom intensity. Dyspnea VAS score ranges from 0 mm (lowest; no dyspnea) to 100 mm (highest; worst dyspnea). Higher scores indicate dyspnea worsening. Baseline measurement was taken before treatment initiation. Per protocol percentage of participants with ≥50% change (percent change calculated: [Week 12 - Baseline]/Baseline*100) and >10 mm absolute change in LCSS-Meso dyspnea score from baseline to Week 12 post treatment initiation is reported here for all randomized participants who had a valid baseline and ≥1 post-baseline value for the LCSS-Meso dyspnea score available.
Time Frame: Baseline, Week 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 299 | 299
Percentage of participants | 15.05 [11.19 to 19.62] | 16.39 [12.38 to 21.08]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p = 0.736, Fisher Exact; Difference in Percentage = -1.3, 95% CI 2-sided [-7.20 to 4.53]

9. Secondary Outcome: Percent Change From Baseline in Forced Vital Capacity (FVC) at Week 12
Description: Pulmonary function test was conducted using a spirometer for assessment of FVC. FVC is the volume of air forcibly exhaled from the lungs after taking the deepest breath possible. Baseline measurement was taken before treatment initiation. Per protocol percent change in FVC from baseline to Week 12 post treatment initiation (percent change calculated: [Week 12 - Baseline]/Baseline*100)] is reported here for all randomized participants who had a valid baseline and ≥1 post-baseline value for FVC available.
Time Frame: Baseline, Week 12
Population: All participants randomized to a study arm who had a valid baseline and ≥1 post-baseline value for FVC available.
Measure: Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 210 | 208
Percent Change | -6.0 [-9.82 to -2.09] | -5.6 [-9.2 to -2.0]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p = 0.979, Longitudinal Model; Difference in Percent Change = -0.06, 95% CI 2-sided [-4.61 to 4.49]

10. Secondary Outcome: Percentage of Participants With ≥10% Change From Baseline in FVC at Week 12
Description: Pulmonary function test was conducted using a spirometer for assessment of FVC. FVC is the volume of air forcibly exhaled from the lungs after taking the deepest breath possible. Baseline measurement was taken before treatment initiation. Per protocol percentage of participants with ≥10% change (percent change calculated: [Week 12 - Baseline]/Baseline*100) in FVC from baseline to Week 12 post treatment initiation is reported here for all randomized participants who had a valid baseline and ≥1 post-baseline value for FVC.
Time Frame: Baseline, Week 12
Population: All participants randomized to a study arm who had a valid baseline and ≥1 post-baseline value for FVC available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 210 | 208
Percentage of participants | 24.76 [19.08 to 31.17] | 21.63 [16.24 to 27.86]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority; p = 0.488, Fisher Exact; Difference in Percentage = 3.1, 95% CI 2-sided [-4.97 to 11.17]

ADVERSE EVENTS:
Time Frame: Up to ~77 months (through database cut-off date of 21-November-2011)
Description: All-Cause Mortality table includes all randomized participants. Serious AEs and other AEs tables include all randomized participants who got ≥1 dose of study drug. Per protocol disease progression of cancer under study was not considered an AE unless it resulted in hospitalization or death. Thus Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Vorinostat | Placebo
All-Cause Mortality (participants affected / at risk) | 288/329 | 284/332
Serious Adverse Events (participants affected / at risk) | 133/329 | 131/329
Other Adverse Events (participants affected / at risk) | 303/329 | 281/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=329) | Placebo (N=329)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (7) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 4 (4)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (14) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Euthanasia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 8 (8) | 2 (2)
General physical health deterioration (General disorders) | 2 (3) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 5 (6) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (3)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 4 (6)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (4)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (15) | 10 (10)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (5) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pleural mesothelioma malignant advanced (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 (51) | 59 (59)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (10)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 25 (28)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=329) | Placebo (N=329)
Anaemia (Blood and lymphatic system disorders) | 45 (86) | 22 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (46) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 28 (32) | 17 (18)
Constipation (Gastrointestinal disorders) | 80 (116) | 69 (96)
Diarrhoea (Gastrointestinal disorders) | 142 (327) | 58 (85)
Dry mouth (Gastrointestinal disorders) | 31 (35) | 17 (23)
Nausea (Gastrointestinal disorders) | 189 (339) | 104 (162)
Vomiting (Gastrointestinal disorders) | 131 (284) | 45 (81)
Fatigue (General disorders) | 153 (277) | 128 (224)
Malaise (General disorders) | 18 (26) | 3 (4)
Oedema peripheral (General disorders) | 23 (26) | 31 (38)
Pyrexia (General disorders) | 38 (54) | 26 (35)
Blood creatinine increased (Investigations) | 29 (35) | 4 (4)
C-reactive protein increased (Investigations) | 19 (22) | 13 (17)
Weight decreased (Investigations) | 67 (97) | 26 (30)
Decreased appetite (Metabolism and nutrition disorders) | 133 (219) | 85 (122)
Dehydration (Metabolism and nutrition disorders) | 19 (23) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (32) | 27 (36)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 (24) | 11 (12)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 59 (79) | 83 (110)
Dizziness (Nervous system disorders) | 23 (39) | 18 (29)
Dysgeusia (Nervous system disorders) | 27 (32) | 19 (20)
Headache (Nervous system disorders) | 23 (89) | 27 (43)
Anxiety (Psychiatric disorders) | 14 (14) | 25 (25)
Insomnia (Psychiatric disorders) | 28 (30) | 23 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 59 (72) | 66 (72)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 97 (139) | 97 (120)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 23 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.